CLINICAL TRIAL: NCT01566552
Title: Point of Care Diagnosis and Treatment With Single Dose Liposomal Amphotericin B for Visceral Leishmaniasis in India.
Brief Title: Single Dose Liposomal Amphotericin B for Visceral Leishmaniasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Banaras Hindu University (Other)
Collaborators: Rajendra Memorial Research Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shyam Sundar, PROFESSOR, Banaras Hindu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHU001/2012
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2012-03

CONDITIONS: Visceral Leishmaniasis
Keywords: AMBISOME; VISCERAL LEISHMANIASIS; SINGLE DOSE
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SINGLE DOSE AMBISOME (Other)
  Interventions: Drug: AMBISOME

INTERVENTIONS:
Drug: AMBISOME — SINGLE DOSE AMBISOME FOR TREATMENT OF VISCERAL LEISHMANIASIS
  Other Names: LIPOSOMAL AMPHOTERECIN B

SUMMARY:
The study is designed to determine the use of delivering point of care, rapid diagnosis with rK39 and treatment with AmBisome single dose of 10 mg/kg when administrated in the Primary Health Center (PHC) settings with regard to operational feasibility, safety and final cure rate at 6 months after end of treatment. Point of care diagnosis and treatment (PCDT) at the PHC level would bring the best available interventions closer to the patients with visceral leishmaniasis (VL) whose villages are within several kilometers of the PHC. This would support the VL elimination program in the Indian subcontinent.

DETAILED DESCRIPTION:
Primary Objectives:

To evaluate the operational feasibility of delivering point of care, rapid diagnosis with rK39 and treatment with AmBisome® single dose of 10 mg/kg, when administrated at the Primary Health Centers (PHC) setting with regard to feasibility and safety .

Secondary objectives:

To determine efficacy of the treatment scheme when delivered by district hospitals and PHC facilities

Methodology:

Three districts, Saran, Simastipur and Muzaffarpur in the VL endemic state of Bihar in India will be selected for the study. Initially, 300 eligible patients will be diagnosed and treated at hospital level with liposomal amphotericin B, using a single dose of 10 mg/kg. If no significant feasibility or safety issues are identified in this group of patients, 1000 additional subjects will be diagnosed and treated at the PHC level. Feasibility will be determined by the proportion of patients attending the PHCs treated with single dose AmBisome and the proportion of patients that need to be referred to the district hospitals for management of adverse events. The initial cure rate will be determined at day 30, after end of treatment (EOT). If initial cure is observed, the patient will be followed up and evaluated 6 months after the end of treatment for final clinical cure.

Study medication, dose and mode of administration Liposomal Amphotericin B (Gilead Sciences, Foster City, CA, USA) is formulated as a lyophilized powder which will be reconstituted in 10 ml of distilled water as a solution and the total dose will be then diluted in three times the volume of 5% dextrose solution.

Total infusion will be done in 2 hours.

Before infusion of AmBisome®, each patient will be given Paracetamol (Adult: 500 mg; Children below 12 years 10 mg/kg) and Chlorpheniramine (Adult: 4mg; Children below 12 years 1-2mg)

Parameters for evaluation Laboratory parameters for safety Adverse event

Endpoints (Feasibility)

* 85% of VL patients attending the PHCs are treated with the single dose AmBisome scheme.
* 3% of patients treated with single dose AmBisome are referred to district hospitals for AEs management .
* 95% of patients treated with single dose AmBisome are cure at 6 months after EOT.

Endpoints (Efficacy) Initial Cure: Defined as remission of fever, any decrease in spleen size compared with baseline, hemoglobin is increased by at least 10% compared to baseline or to at least 10g/dl, and improvement in other clinical signs and symptoms on day 30.

Final Cure: Defined on the fulfillment of following criteria at 6 months after EOT: No relapse after initial cure, absence of fever and no increase in spleen size compared with day 30 and hemoglobin is increased by at least10% compared to day 30 or to at least 10g/dl.

Statistical methods Efficacy analysis: Calculation of cure rate with 95% and 90% lower confidence limit according to the Clopper Pearson method.

Safety analysis: Calculation of overall incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 5 years of age
2. History of fever for more than 2 weeks
3. Splenomegaly
4. rK 39 rapid test positive
5. Biochemical and hematological test values as follows:

   * Hemoglobin ≥ 5 g/dl
   * White blood cell count ≥1.0 x 109/L
   * AST, ALT ≤ 3 times the upper limit of normal
   * Serum creatinine level within normal limit
6. Written informed consent from the patient/ or parent or guardian if under 18 years old.

Exclusion Criteria:

1. A history of intercurrent or presence of clinical signs / symptoms of concurrent diseases / conditions (e.g. Chronic alcohol consumption or drug addiction, renal, hepatic, cardiovascular or CNS disease; diabetes mellitus, dehydration, other infectious diseases or major psychiatric diseases) only if the intercurrent conditions are not under control before starting the treatment with AmBisome.
2. Any condition which according to the investigator might prevent the patient from completing the study therapy and subsequent follow up
3. A history of allergy or hypersensitivity to Amphotericin B
4. Previous treatment for VL
5. Prior treatment failure with Amphotericin B
6. Post Kala-azar Dermal Leishmaniasis (PKDL

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
CLINICAL CURE | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: SHYAM SUNDAR, M.D., Principal Investigator — Banaras Hindu University
Locations (1):
- Kala Azar Medical Research Center, Muzaffarpur, Bihar, India